CLINICAL TRIAL: NCT03255928
Title: Analysis of the Platelet Activity State in Patients Implanted With Ventricular Assist Device (VAD)
Brief Title: Dynamics of Platelet Activation in Patients With Ventricular Assist Device (VAD)
Acronym: PASVAD
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Collaborators: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Filippo Consolo, Assistant Professor, Scientific Institute San Raffaele
Other Study IDs: PASVAD v. n°1 10/03/2017
Record Dates: First submitted 2017-07-28; First posted 2017-08-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Thrombosis; Blood Coagulation Disorder; Platelet Thrombus; Platelet Dysfunction Due to Aspirin; Failure;Ventricular
Keywords: Platelet activation; Ventricular Assist Device; Thrombosis; Bleeding; Antithrombotic Pharmacological Therapy; Mechanical Circulatory Support
MeSH Terms: conditions — Thrombosis; Blood Coagulation Disorders; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Platelet-free-plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- VAD-implanted patients: All patients receiving a VAD implant
  Interventions: Diagnostic Test: PAS assay, TGT
- VAD-patients suffering adverse events (AE): VAD-patients sustaining a thromboembolic/bleeding complication over the course of support
  Interventions: Diagnostic Test: PAS assay, TGT

INTERVENTIONS:
Diagnostic Test: PAS assay, TGT — Evaluation of platelet function

SUMMARY:
Consenting patients with end-stage heart failure that are implanted with/candidates for implant of a short-term/durable mechanical circulatory support device (e.g.: percutaneous microaxial pumps (Impella), extracorporeal membrane oxygenator (ECMO), Ventricular Assist Device (VAD) will be enrolled in the study.

Aim of the study is to evaluate the patients' haemostatic and coagulation profile, how it interacts with the support device as well as the effect of antithrombotic drugs. From these data, it will be possible to derive the mechanisms triggering post-implant thromboembolic/hemorrhagic complications and to identify potential therapeutic targets.

DETAILED DESCRIPTION:
The study is aimed at evaluating the patients' haemostatic and coagulation profile focusing, in particular, on platelet function. Platelet function will be analyzed utilizing two innovative analytic diagnostic tests, namely i) the Platelet Activity State (PAS) assay and ii) the Thrombin Generation Test (TGT).

PAS values and TGT will be measured at different time-points over the course of support:

i) before the implant of the support system, to define baseline patients' characteristics; ii) in the early-post implant, during patient hospitalization; iii) during long-term follow up, to evaluate the dynamics of platelet function over the course of support and potential alterations of platelet-mediated haemostatic processes; iv) at the occurrence of any thromboembolic/hemorrhagic complication or following a modification of the antithrombotic pharmacological therapy.

Platelet function will be evaluated through:

i) the Platelet Activity State (PAS) assay, a biochemical assay able to quantify the platelet thrombin production rate and to correlate this rate with the actual level of platelet activation (i.e., the platelet pro-thrombotic tendency); ii) the Thrombin Generation Test (TGT), a biochemical assay that the investigators have properly modified to account selectively for the platelet contribution on plasmatic thrombin generation.

PAS and TGT experimental values will be correlated with the occurrences of post-implant complications. Experimental values will be also correlated with standard clinical parameters of coagulation and hemolysis, such as: platelet count, hematocrit, hemoglobin, prothrombin time (PT), activated partial thromboplastin time (aPTT), International Normalized Ratio (INR), D-Dimer, Fibrinogen, L-lactate dehydrogenase, haptoglobin, plasma-free hemoglobin, and C-reactive protein levels. Also levels of thrombin-antithrombin complex, Von Willebrand factor, prothrombin1,2 fraction and tissue factor, will be measured and recorded. In addition, pump (i.e. VAD) working parameters (i.e., rotation velocity, cardiac outflow and power consumption) will be recorded. Log-files of the pump will be downloaded and analyzed to characterize the correlation with the development of adverse events (AV). Finally, antithrombotic therapy will be recorded and used in the study.

ELIGIBILITY:
Inclusion Criteria:

* All consenting patients candidates for short-term (Impella, ECMO) or durable (LVAD) mechanical circulatory support device implantation
* All consenting patients that are implanted with short-term (Impella, ECMO) or durable (LVAD) mechanical circulatory support device

Exclusion Criteria:

- Patients < 18-years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with end-stage heart failure receiving a mechanical circulatory support system
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events. Change of PAS assay from baseline to 24 months post-implant | Through study completion. Specific time-points: 1, 3, 6, 12, 18, and 24 months post-implant and at the occurrence of any AE
  Correlation between platelet activation and the development of post-implant complications
Number of participants with treatment-related adverse events. Change of TGT from baseline to 24-months post-implant | Through study completion. Specific time-points: 1, 3, 6, 12, 18, and 24 months post-implant and at the occurrence of any AE
  Correlation between platelet pro-thrombinase activity and the development of post-implant complications
Number of participants with treatment-related adverse events. Change of clinical and coagulation parameters from baseline to 24-months post-implant | Through study completion. Specific time-points: 1, 3, 6, 12, 18, and 24 months post-implant and at the occurrence of any AE
  Correlation between coagulation parameters and the development of post-implant complications
Number of participants with treatment-related adverse events. Change of pump working conditions after the device implant | Through study completion. Specific time-points: 1, 3, 6, 12, 18, and 24 months post-implant and at the occurrence of any AE
  Correlation between pump working conditions and the development of post-implant complications

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events. Change of prescribed antithrombotic therapy (anticoagulation and antiplatelet drugs) from baseline to 24 months post-implant | Through study completion. Specific time-points: 1, 3, 6, 12, 18, and 24 months post-implant and at the occurrence of any AE
  Correlation between antithrombotic therapy and the development of post-implant complications

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Consolo, PhD, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientifc Institute - Cardiothoracic Intensive Care Unit, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
Privacy restrictions

REFERENCES:
- [Background] Valerio L, Consolo F, Bluestein D, Tran P, Slepian M, Redaelli A, Pappalardo F. Shear-mediated platelet activation in patients implanted with continuous flow LVADs: A preliminary study utilizing the platelet activity state (PAS) assay. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:1255-8. doi: 10.1109/EMBC.2015.7318595. PMID 26736495
- [Background] Consolo F, Sheriff J, Gorla S, Magri N, Bluestein D, Pappalardo F, Slepian MJ, Fiore GB, Redaelli A. High Frequency Components of Hemodynamic Shear Stress Profiles are a Major Determinant of Shear-Mediated Platelet Activation in Therapeutic Blood Recirculating Devices. Sci Rep. 2017 Jul 10;7(1):4994. doi: 10.1038/s41598-017-05130-5. PMID 28694489
- [Background] Sheriff J, Girdhar G, Chiu WC, Jesty J, Slepian MJ, Bluestein D. Comparative efficacy of in vitro and in vivo metabolized aspirin in the DeBakey ventricular assist device. J Thromb Thrombolysis. 2014 May;37(4):499-506. doi: 10.1007/s11239-013-0997-6. PMID 24043375
- [Background] Sheriff J, Bluestein D, Girdhar G, Jesty J. High-shear stress sensitizes platelets to subsequent low-shear conditions. Ann Biomed Eng. 2010 Apr;38(4):1442-50. doi: 10.1007/s10439-010-9936-2. Epub 2010 Feb 5. PMID 20135353
- [Background] Jesty J, Bluestein D. Acetylated prothrombin as a substrate in the measurement of the procoagulant activity of platelets: elimination of the feedback activation of platelets by thrombin. Anal Biochem. 1999 Jul 15;272(1):64-70. doi: 10.1006/abio.1999.4148. PMID 10405294
- [Background] Slepian MJ, Sheriff J, Hutchinson M, Tran P, Bajaj N, Garcia JGN, Scott Saavedra S, Bluestein D. Shear-mediated platelet activation in the free flow: Perspectives on the emerging spectrum of cell mechanobiological mechanisms mediating cardiovascular implant thrombosis. J Biomech. 2017 Jan 4;50:20-25. doi: 10.1016/j.jbiomech.2016.11.016. Epub 2016 Nov 10. PMID 27887727
- [Background] Rogers JG, Pagani FD, Tatooles AJ, Bhat G, Slaughter MS, Birks EJ, Boyce SW, Najjar SS, Jeevanandam V, Anderson AS, Gregoric ID, Mallidi H, Leadley K, Aaronson KD, Frazier OH, Milano CA. Intrapericardial Left Ventricular Assist Device for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):451-460. doi: 10.1056/NEJMoa1602954. PMID 28146651
- [Background] Slaughter MS, Pagani FD, McGee EC, Birks EJ, Cotts WG, Gregoric I, Howard Frazier O, Icenogle T, Najjar SS, Boyce SW, Acker MA, John R, Hathaway DR, Najarian KB, Aaronson KD; HeartWare Bridge to Transplant ADVANCE Trial Investigators. HeartWare ventricular assist system for bridge to transplant: combined results of the bridge to transplant and continued access protocol trial. J Heart Lung Transplant. 2013 Jul;32(7):675-83. doi: 10.1016/j.healun.2013.04.004. PMID 23796152
- [Background] Valerio L, Tran PL, Sheriff J, Brengle W, Ghosh R, Chiu WC, Redaelli A, Fiore GB, Pappalardo F, Bluestein D, Slepian MJ. Aspirin has limited ability to modulate shear-mediated platelet activation associated with elevated shear stress of ventricular assist devices. Thromb Res. 2016 Apr;140:110-117. doi: 10.1016/j.thromres.2016.01.026. Epub 2016 Feb 1. PMID 26938158
- [Background] Consolo F, Sferrazza G, Motolone G, Contri R, Valerio L, Lembo R, Pozzi L, Della Valle P, De Bonis M, Zangrillo A, Fiore GB, Redaelli A, Slepian MJ, Pappalardo F. Platelet activation is a preoperative risk factor for the development of thromboembolic complications in patients with continuous-flow left ventricular assist device. Eur J Heart Fail. 2018 Apr;20(4):792-800. doi: 10.1002/ejhf.1113. Epub 2017 Dec 28. PMID 29282819
- [Background] Consolo F, Pozzi L, Sferrazza G, Della Valle P, D'Angelo A, Slepian MJ, Pappalardo F. Which Antiplatelet Therapy in Patients With Left Ventricular Assist Device and Aspirin Allergy? Ann Thorac Surg. 2018 Feb;105(2):e47-e49. doi: 10.1016/j.athoracsur.2017.09.022. PMID 29362190
- [Background] Consolo F, Sferrazza G, Motolone G, Pieri M, De Bonis M, Zangrillo A, Redaelli A, Slepian MJ, Pappalardo F. Shear-Mediated Platelet Activation Enhances Thrombotic Complications in Patients With LVADs and Is Reversed After Heart Transplantation. ASAIO J. 2019 May/Jun;65(4):e33-e35. doi: 10.1097/MAT.0000000000000842. PMID 29952802
- [Derived] Foglieni C, Ravanelli D, Lombardi M, Spartano L, Pieri M, Ajello S, Landoni G, Scandroglio AM, Consolo F. Platelet microRNA Expression Can Predict Bleeding in HeartMate3 Patients Treated With or Without Aspirin. J Cardiovasc Transl Res. 2025 Oct;18(5):1032-1041. doi: 10.1007/s12265-025-10659-2. Epub 2025 Jul 11. PMID 40643853
- [Derived] Consolo F, Pieri M, Pazzanese V, Scandroglio AM, Pappalardo F. Longitudinal analysis of pump parameters over long-term support with the HeartMate 3 left ventricular assist device. J Cardiovasc Med (Hagerstown). 2023 Oct 1;24(10):771-775. doi: 10.2459/JCM.0000000000001522. Epub 2023 Jun 30. PMID 37409664
- [Derived] Consolo F, Marasi A, Della Valle P, Bonora M, Pieri M, Scandroglio AM, Redaelli A, Zangrillo A, D'Angelo A, Pappalardo F. Bleeding in patients with continuous-flow left ventricular assist devices: acquired von Willebrand disease or antithrombotics? Eur J Cardiothorac Surg. 2022 Jun 15;62(1):ezab474. doi: 10.1093/ejcts/ezab474. PMID 34718493
- [Derived] Consolo F, Pappalardo F. Real-Time Analysis of the Log Files of the HeartWare Continuous-Flow Left Ventricular Assist Device for the Early Diagnosis of Pump Thrombosis: a Step Forward Toward Clinical Translation. J Cardiovasc Transl Res. 2022 Apr;15(2):408-415. doi: 10.1007/s12265-021-10157-1. Epub 2021 Jul 19. PMID 34282539